CLINICAL TRIAL: NCT04374422
Title: Effect of SARS- COVID-19 Pandemic on Female Sexual Behavior
Brief Title: COVID-19 Pandemic and Female Sexual Behavior
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: AcibademU cov
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Sexual Behavior; COVID
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: study group pre-pandemic time interval
  Interventions: Behavioral: fsfi survey
- 2: same population during pandemic
  Interventions: Behavioral: fsfi survey

INTERVENTIONS:
Behavioral: fsfi survey — sexual behavior Questionaire

SUMMARY:
World Health Organization declared new SARS-CoV-2 infection a pandemic, and many states enacted strict, rules such as border closures, transportation restrictions and quarantine.Many studies in the literature have described the relationship between mass disasters and female sexual behavior, but none have investigated the effect of SARS-CoV-2 pandemic on women's sexual attitude. The aim of this study is therefore to evaluate the effect of SARS-CoV-2 pandemic on female sexual behavior.

DETAILED DESCRIPTION:
Coronaviruses are a group of RNA viruses that affect mainly the respiratory system and cause the common cold, fever, and coughs in mammals and birds. However, in some cases, coronaviruses are associated with more serious and lethal conditions, such as pneumonia, bronchitis, and severe acute respiratory syndrome. A novel coronavirus (SARS-CoV-2) originating from Wuhan, China led to a global health crisis. At the time of writing, SARS-CoV-2 infected more than two million, resulting in almost 180.000 deaths. World Health Organization declared new SARS-CoV-2 infection a pandemic, and many states enacted strict, rules such as border closures, transportation restrictions, and quarantine.

The term 'sexual behavior' encompasses a large spectrum of actions in which humans present their sexuality. Previous reports have analyzed the effect of mass disasters on female sexual behavior.

Many studies in the literature have described the relationship between mass disasters and female sexual behavior, but none have investigated the effect of the SARS-CoV-2 pandemic on women's sexual attitude. The aim of this study is therefore to evaluate the effect of the SARS-CoV-2 pandemic on female sexual behavior.

ELIGIBILITY:
Inclusion Criteria:

* married
* above 18 yo
* premenopausal status

Exclusion Criteria:

* urinary incontinence
* history of gynecologic operation
* malignancy
* psychiatric or neurologic disease diagnosis
* being infected by HBV HCV or HIV

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female sexual function
Study Population: From February 2018 to September 2019. For each participant, detailed medical history was obtained, including age, body mass index (BMI), education and income level, presence of comorbidities and the number of previous deliveries. Other details noted were menstrual status of patients, frequency of sexual intercourse and desire for fertility. All patients were asked to fill out the Female Sexual Function Index (FSFI) form. Patients' data were recorded in the electronic data system, prospectively.
  To identify the effect of SARS-CoV-2 pandemic on female sexual behavior, the investigators conducted an observational study to compare the frequency of sexual intercourse, desire for fertility, FSFI score, contraception type and presence of vaginal infection between pandemic era (March 11th and April 12th 2020) and 6-12 months prior to the pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-04-12 (Actual); Study Completion 2020-04-12 (Actual)

PRIMARY OUTCOMES:
FSFI (Female Sexual Function Index)SCORE difference | 1 year
  the FSFI SCORE difference between pre and during pandemic

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
in case of request

REFERENCES:
- [Result] Liao X, Wang B, Kang Y. Novel coronavirus infection during the 2019-2020 epidemic: preparing intensive care units-the experience in Sichuan Province, China. Intensive Care Med. 2020 Feb;46(2):357-360. doi: 10.1007/s00134-020-05954-2. Epub 2020 Feb 5. No abstract available. PMID 32025779
- [Result] Liu S, Han J, Xiao D, Ma C, Chen B. A report on the reproductive health of women after the massive 2008 Wenchuan earthquake. Int J Gynaecol Obstet. 2010 Feb;108(2):161-4. doi: 10.1016/j.ijgo.2009.08.030. Epub 2009 Nov 4. PMID 19892335